CLINICAL TRIAL: NCT03225573
Title: The Prevalence of a Second Mesiobuccal Canal of Maxillary First and Second Molars Using CBCT Among Egyptian Population: A Cross-Sectional Study
Brief Title: Prevalence of Second Mesiobuccal Canal of Maxillary First and Second Molars Among Egyptian Population
Acronym: CBCT
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Prof. Nashwa Salah, Professor of Oral and Maxillofacial Radiology Faculty of Dentistry, Cairo University
Other Study IDs: Rad2:5:1
Record Dates: First submitted 2017-07-11; First posted 2017-07-21 (Actual); Results first posted 2020-02-11 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Second Mesiobuccal Canal; Maxillary First and Second Molars
Keywords: second mesiobuccal canal CBCT prevalence population

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
a cross-sectional study to estimate the prevalence of a second mesiobuccal canal of maxillary first and second molars in Egyptian population using cone beam computed tomography through retrospective data analysis

DETAILED DESCRIPTION:
Setting and Location:

1. The data collection will be obtained from the data base available at a private radiographic centre ORASCAN Oral & Maxillofacial Imaging Centre located in Cairo, Egypt.
2. CBCT images will be obtained from Egyptian patients who had CBCT examination as part of their dental examination, diagnosis or treatment planning during the years 2015-16-17.

Participants:

A total of 196 CBCT scans of Maxillary first and second permanent molars belonging to Egyptian individuals will be included.

Variables:

1. Number of root canals in mesiobuccal root of first and second maxillary molars
2. Sex of the patient will be identified and addressed as the prevalence of the second mesiobuccal canal may show sex predilection

Data Sources / Measurements:

Retrospective Data Analysis will be performed after the CBCT images are pooled from the computer database.

All the CBCT examinations were scanned using Cranex® 3D SOREDEX, 0.2 voxel resolution, 8 × 6 cm FOV, 90 kVp, 10 mA and 6 seconds exposure time.

CBCT images will be analysed in the 3 planes; first the sagittal and coronal sections will be oriented parallel to the long axis of the root, and then sections will be obtained on the axial plane for detection of the 2nd mesiobuccal canal.

CBCT images will be interpreted by three oral radiologists independently; blinded from demographic data of the patients and from the results of each other.

Each one will evaluate the images separately twice with a period of two weeks between the two reading sessions.

Then inter-observational and intra-observational variability between the observers will be evaluated.

The sex of the patient will be identified from the patient's demographic data available on the patient's file on the database of the private radiographic centre.

Bias:

No source of bias.

Study Size:

The aim of the study is to assess the prevalence of a second mesiobuccal canal of maxillary first and second molars in Egyptian population. Based on the previous paper by Nikoloudaki et al, 2015, the prevalence of Second Mesiobuccal Canal of Maxillary First and Second Molars was 89 and 85%. Using a precision of 5, a design effect set at 1 with 95% CI (confidence interval), a total sample size of 196 will be sufficient. The sample size was calculated by Epi info.

Sampling Strategy: The sample will be collected by simple random sampling.

Quantitative Variables:

The number of CBCT scans of Egyptian individuals with second mesiobuccal canal will be counted to estimate the prevalence of the second mesiobuccal canal.

Statistical Methods:

1. Data will be analysed using IBM SPSS advanced statistics (Statistical Package for Social Sciences), version 21 (SPSS Inc., Chicago, IL). Numerical data will be described as mean and standard deviation or median and range. Categorical data will be described as numbers and percentages. Comparisons between male and females for normally distributed numeric variables will be done using the Student's t-test while for non-normally distributed numeric variables will be done by Mann-Whitney test. Comparisons between categorical variables will be performed using the chi square test. A p-value less than or equal to 0.05 will be considered statistically significant. All tests will be two tailed.
2. If the patient's age couldn't be found in the patient's file, the dental age will be used.
3. If the patient's sex couldn't be found in the patient's file, the patient's name will be used to indicate the sex. Patients with mixed name will be excluded.

ELIGIBILITY:
Inclusion Criteria:

* First and second maxillary permanent molars of Egyptian patients starting from 15 years, males or females
* Intact roots without fractures or cracks
* Molars without posts or previous root canal treatment
* CBCT scans of maxillary first and second molars using 8 × 6 Field of view, 0.2 voxel resolution

Exclusion Criteria:

* Evidence of apicectomy or periapical surgery
* Odontogenic or non-odontogenic pathology
* Maxillary molars with developmental anomalies
* External or Internal Root resorption
* Canal Calcification
* Previous root canal treatment
* Extensive coronal restorations
* Posts or crown restorations
* Root caries specially reaching the trifurcation area
* Tomographic images of poor quality or artifacts interfering with the detection of root canals

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Egyptian Population
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-04-15 (Actual); Study Completion 2018-05-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- ORASCAN Oral and Maxillofacial Imaging Centre, Cairo, Maadi, Egypt

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: molar teeth
Groups:
- Egyptian Patients: Egyptian patients who had CBCT examination as part of their dental examination, diagnosis or treatment planning during the years 2015-16-17.
  starting from 15 years, males or females
Period: Overall Study
Arm/Group | Egyptian Patients
Started | 60; 198 molar teeth
Completed | 60; 198 molar teeth
Not Completed | 0; 0 molar teeth

BASELINE CHARACTERISTICS:
Units Other Than Participants: molar teeth
Arm/Group | Egyptian Patients
Number analyzed (Participants) | 60
Number analyzed (molar teeth) | 198
Age, Categorical [Count of Units; unit: molar teeth] — Population: the number analyzed is the total number of molar teeth (198) analyzed from the 60 scans of the patients
  molar teeth
    <=18 years | 0
    Between 18 and 65 years | 198
    >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — race and ethnicity not collected
  Participants
    Hispanic or Latino | 0
    Not Hispanic or Latino | 0
    Unknown or Not Reported | 60
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 60
Region of Enrollment [Number; unit: molar teeth]
  Egypt | 198

OUTCOME MEASURES:

1. Primary Outcome: Number of Maxillary Molars With a Second Mesiobuccal Canal
Description: measuring device is CBCT software On Demand 3D® , measuring unit is binary system (yes/no)
Time Frame: 1 month
Measure: Count of Units; unit: molar teeth
Units Other Than Participants: molar teeth
Arm/Group | Egyptian Patients
Number analyzed (Participants) | 60
Number analyzed (molar teeth) | 198
molar teeth | 86

ADVERSE EVENTS:
Description: all-cause mortality, serious and other adverse events were not monitored/assessed
Arm/Group | Egyptian Patients
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-06): https://cdn.clinicaltrials.gov/large-docs/73/NCT03225573/Prot_SAP_001.pdf